CLINICAL TRIAL: NCT00436228
Title: An Open-Label, Randomized, Crossover Study to Estimate the Formulation Effect on the Relative Bioavailability of Single Dose Oral SB-742510 in Healthy Subjects
Brief Title: To Study And Compare Bioavailability And Safety Of Four Different Formulations Of The Study Drug
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: OPB107935
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Healthy Subjects
Keywords: healthy volunteer,; Bioavailability,; safety; Phase I,

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
SB-742510 is a semi-synthetic pleuromutilin antibiotic that is being developed for treatment of respiratory infections.

The purpose of this study is to estimate the bioavailability of four different formulations and to evaluate the safety of each of the four formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on medical evaluations performed at screening.
* Healthy adults between 18 and 60 years of age, inclusive.
* Body weight proportional to height.
* Capable of giving written informed consent.
* Female subjects must be of non-childbearing potential.
* QTc less than 450 msec at screening

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history and physical or on the 12-lead surface electrocardiogram at screening or pre-dose.
* The subject has a positive pre-study alcohol/urine drug screen.
* History of regular use of tobacco, or nicotine-containing products.
* A positive pre-study HIV antibody, Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody result within 3 months of screening.
* Use of certain prescription or non-prescription drugs, including vitamins, herbal and dietary supplements.
* An unwillingness to comply with lifestyle and/or dietary restrictions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States